CLINICAL TRIAL: NCT03194347
Title: Clinical Value of Molecular Genetic Analyzes in Gynecological Malignomas
Acronym: MAGynMA
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: MAGynMA
Record Dates: First submitted 2017-05-22; First posted 2017-06-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Gynecologic Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: molecular genetic analyses — molecular genetic analyses

SUMMARY:
The aim of the planned research project is to find out the clinical significance of molecular genetic analyzes in gynecological malignomas. In particular, it will be investigated how the knowledge of a molecular-genetic finding affects the therapeutic decision of the physician. Furthermore, genetic changes in the tumor tissue will be compared with the changes in CTCs, DTCs and cfDNA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a solid tumor disease
* The presence of a molecular genetic diagnosis of the tumor tissue from practice for human genetics
* Age > 18 years
* informed consent

Exclusion Criteria:

* life expectancy <12 months or worse general condition (Karnofsky <70)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — gynecological tumors
Study Population: All patients with a gynecological malignancy, in whom a genetic testing of tumor tissue (somatic mutation) and blood cells (germ line mutation) has already taken place.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of molecular genetic findings to the therapy decision | 3years
  It will be analyzed if the physicians selection of a therapy is influenced by a present molecular genetic finding. Therapy recommondation based on molecular genetic analysis will be compared with the acutal therapy decision.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas D Hartkopf, Prof, Principal Investigator — Department of Women's Health
Locations (1):
- University Women's Hospital, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No